CLINICAL TRIAL: NCT06618625
Title: The Effect of Tube Rotation on Passage of Tracheal Tube Through Nasopharynx Into the Oral Cavity in Nasotracheal Intubation
Brief Title: Tube Rotation for Tube Passage Into the Oral Cavity in Nasotracheal Intubation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 10-2023-61
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Nasotracheal Intubation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rotation (Experimental): For nasotracheal intubation, the nasal RAE tube will be inserted with it rotated by 90 degrees in counter-clockwise direction for patients in the 'Rotation' arm.
  Interventions: Procedure: nasotracheal intubation
- Neutral (Active Comparator): For nasotracheal intubation, the nasal RAE tube will be inserted without tube rotation for patients in the 'Neutral' arm.
  Interventions: Procedure: nasotracheal intubation

INTERVENTIONS:
Procedure: nasotracheal intubation — For nasotracheal intubation, the nasal RAE tube will be inserted with it rotated by 90 degrees in counter-clockwise direction for patients in the 'Rotation' arm.
  For nasotracheal intubation, the nasal RAE tube will be inserted without tube rotation for patients in the 'Neutral' arm.

SUMMARY:
The purpose of the study is to investigate the effect of tube rotation on passage of the tracheal tube through the nasopharynx into the oral cavity in nasotracheal intubation.

DETAILED DESCRIPTION:
This prospective randomized controlled study was approved by IRB of our institute.

Patients requiring nasotracheal intubation will be screened for eligibility of the study. Then, patients will be randomized to one of two groups; (group I: tube advancement in neutral / group II: tube advancement with the tube counter-clockwise rotated). After induction of anesthesia and muscle relaxation, the preformed nasal RAE (Ring-Adair-Elwyn) tube will be inserted via a nostril approximately 3-4 cm. Next, an anesthesiologist will advance the tube, with it neutral, continuously into the oral cavity of the patients in Group I, while the anesthesiologist will advance the tube, with it rotated counter-clockwise in 90 degree, into the oral cavity of the patients in Group II. After the tube will be placed in the oral cavity, the anesthesiologist will perform nasotracheal intubation with Magill forceps. After that, an investigator will check occurrence of epistaxis due to nasotracheal intubation and its severity with a fiberoptic bronchoscope. After obtainment of all data, investigators will analyze incidence of epistaxis and its severity between two groups.

ELIGIBILITY:
Inclusion Criteria:

* adult patients requiring nasotracheal intubation for elective surgery

Exclusion Criteria:

* refuse to participate in the study
* severe deformity in nose
* current severe epistaxis
* limitation of neck extension

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-23 (Estimated); Primary Completion 2025-08-22 (Estimated); Study Completion 2025-09-22 (Estimated)

PRIMARY OUTCOMES:
tube blockade | during tube advancement from the nasal cavity to the oral cavity
  tube blockade when an anesthesiologist is advancing the tracheal tube from the nasal cavity to the oral cavity.

SECONDARY OUTCOMES:
epistaxis | during nasotracheal intubation
  epistaxis due to nasotracheal intubation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim H, Lee JM, Lee J, Hwang JY, Chang JE, No HJ, Won D, Row HS, Min SW. Effect of neck extension on the advancement of tracheal tubes from the nasal cavity to the oropharynx in nasotracheal intubation: a randomized controlled trial. BMC Anesthesiol. 2019 Aug 17;19(1):158. doi: 10.1186/s12871-019-0831-6. PMID 31421677